CLINICAL TRIAL: NCT02155075
Title: Evaluation of Real Imaging's 3d Functional Metabolic Imaging and Risk Assessment (Mira) System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 960-CSP-ISR_ImplantsMC_ILS3
Record Dates: First submitted 2014-06-01; First posted 2014-06-04 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Breast neoplasm; Breast implants; Mammography; Breast imaging; Imaging augmented breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Testing phase (Phase II) Arm 1 - 180 participant will be enrolled for this arm. Participants will be enrolled to undergo MIRA device imaging. Following the MIRA device imaging procedure, the optimized risk model will assign a binary result to the participant.
  All participants will recive standart of care, participants with negative screening exams and a positive MIRA device imaging result will additionally undergo MRI.
  Interventions: Device: MIRA device imaging
- Arm 2 (Experimental): Testing phase (Phase II) Arm 2 - 150 participant will be enrolled for this arm. Participants will be enrolled to undergo MIRA device imaging. Following the MIRA device imaging procedure all participants in arm 2 will be following standard of care, MIRA device imaging will NOT change their clinical path.
  Interventions: Device: MIRA device imaging

INTERVENTIONS:
Device: MIRA device imaging — MIRA device imaging for adjunctive detection of breast cancer. Arm 1 administarte result
  Other Names: Real imager 8 (RI8)

SUMMARY:
Three-dimensional functional Metabolic Imaging (3D MIRA) is a new infrared imaging technology using the Real Imager 8 (RI8) developed by Real Imaging. This technology generates 3D metabolic maps of the breast and based on sophisticated machine learning technology, provides objective risk assessment for the presence of malignant tumor in the breast. The procedure is non-invasive, comfortable and does not involve ionizing radiation. It is based on acquiring infrared images of the breast. Those images are processed and analyzed by computers to provide the objective risk assessment.

The technology is intended to be used as a screening tool for breast cancer and emerges as highly useful in women for whom screening mammography is sub-optimal, such as women with dense breast. 3D MIRA is unaffected by breast density and is therefore ideal for evaluating patients with mammographically dense breasts.

The purpose of this clinical study is to assess the ability of this novel technology to detect breast cancer in women.

ELIGIBILITY:
PHASE 1:

INCLUSION CRITERIA

1. Female
2. Woman has read, understood and signed the inform consent form
3. Age: 30 years and older
4. A. Women who are scheduled to undergo routine Mammography and/or US and/or MRI screening OR B. Women summoned for breast biopsy following a suspicious finding in recent screening exam and was graded 4/5 on BI-RADS scale

EXCLUSION CRITERIA:

1. Women who have had a Mammography and/or US and/or MRI examination performed on the day of the study prior to MIRA scan
2. Women who had undergone mastectomy and/or breast reconstruction
3. Women who have had a breast biopsy performed throughout the 6 weeks preceding the study
4. Women who have a fever on the day of the MIRA imaging
5. Women who are pregnant
6. Women who are breast-feeding
7. Women with implanted pacemaker/defibrillator, implanted venous access device (portacath) or other implanted devices in the chest area
8. Women who are unable to read, understand and execute written informed consent
9. Women who are currently undergoing chemotherapy and/or radiotherapy

PHASE 2:

ARM 1:

INCLUSION CRITERIA

1. Female
2. Age: 30 years and older
3. A. Asymptomatic women who are scheduled to undergo routine screening mammography or routine screening mammography and US Or B. Subjects scheduled for image-guided needle biopsy as a result of findings obtained during standard of care imaging modalities (mammography, ultrasound and/or MRI).

5. Women whose most recent prior mammogram was interpreted as heterogeneously dense (ACR BI-RADS Breast Density C) or extremely dense (ACR BI-RADS Breast Density D).

EXCLUSION CRITERIA:

1. Subjects who have had a Mammography and/or US and/or MRI examination performed on the day of the study prior to MIRA scan
2. Subjects scheduled for a diagnostic mammography due to a suspicious lump
3. Subjects who had undergone mastectomy and/or breast reconstruction
4. Subjects who have undergone breast reduction or breast augmentation.
5. Subjects who have large breast scar / breast deformation.
6. Subjects who have significant existing breast trauma.
7. Subjects who have undergone lumpectomy
8. Subjects who have had a breast needle biopsy performed throughout the 6 weeks preceding the study
9. Subjects with implanted pacemaker/defibrillator, implanted venous access device (portacath) or other implanted devices in the chest area
10. Subjects with known Raynaud's Disease.
11. Subjects who have a fever on the day of the MIRA imaging
12. Subjects who are pregnant
13. Subjects who are breast-feeding
14. Subjects with known Mastitis
15. Subjects who are currently undergoing chemotherapy and/or radiotherapy
16. Subjects with contraindication to bilateral mammography or MRI.
17. Subjects who participated in the Calibration Phase will not be able to participate in the Testing Phase.
18. Subjects currently participating in another clinical study.
19. Subjects who are unable to read, understand and execute written informed consent

ARM 2:

INCLUSION CRITERIA:

1. Female
2. Age: 30 years and older
3. Asymptomatic women who are scheduled to undergo routine screening mammography or routine screening mammography and US

EXCLUSION CRITERIA :

1. Subjects who have had a Mammography examination performed on the day of the study prior to MIRA scan
2. Subjects scheduled for a diagnostic mammography due to a suspicious lump
3. Subjects who have had a breast biopsy performed throughout the 6 weeks preceding the study
4. Subjects who have a fever on the day of the MIRA imaging
5. Subjects who are pregnant
6. Subjects who are breast-feeding
7. Subjects with known Mastitis
8. Subjects with known Raynaud's Disease.
9. Subjects who are currently undergoing chemotherapy and/or radiotherapy
10. Subjects with contraindication to bilateral mammography
11. Subjects who participated in the Calibration Phase will not be able to participate in the Testing Phase.
12. Subjects currently participating in another clinical study.
13. Subjects who are unable to read, understand and execute written informed consent

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Sufficient number of cancer case and controls have been imaged | up to 24 months
  As this is a data collection study, end point will be reached when approximately 50 women with breast cancer and 100 healthy women (controls) are imaged by the device and sufficient for the comparison statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Miri Sklair-Levy, MD, Principal Investigator — The Chaim Sheba Medical center at Tel-Hashomer
Locations (1):
- The Chaim Sheba Medical Center at Tel Hashomer, Ramat Gan, Israel